CLINICAL TRIAL: NCT06764368
Title: A Phase II, Single-arm, Multicenter Clinical Study of Adebrelimab Combined With Chemotherapy and Apatinib as First-line Treatment for Unresectable Locally Advanced or Metastatic Pulmonary Neuroendocrine Tumors
Brief Title: Phase II Study of Adebrelimab, Chemotherapy, and Apatinib for Advanced Pulmonary Neuroendocrine Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Chest Hospital (Other)
Responsible Party: Principal Investigator, Tongmei Zhang, Chief Physician, Associate Professor, MD, Beijing Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XKZH-2024-01R
Record Dates: First submitted 2024-12-23; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subtype 1/2/3 (Experimental)
  Interventions: Drug: Adebrelimab + Apatinib

INTERVENTIONS:
Drug: Adebrelimab + Apatinib — Induction Phase:
  Subjects will receive Adebrelimab (1200 mg, Day 1) + Etoposide (100 mg/m2, Days 1-3) + Carboplatin (AUC = 4-5, Day 1) / Cisplatin (75 mg/m2, Day 1) (as determined by the investigator) + Apatinib (250 mg, orally, once daily) in 3-week cycles (Q3W) for 4 to 6 cycles.
  Maintenance Phase:
  Adebrelimab (1200 mg, Day 1) + Apatinib (250 mg, orally, once daily) will be administered for 1 year or until one of the following occurs: disease progression, intolerable toxicity, withdrawal of informed consent by the subject, voluntary withdrawal from the study, or other protocol-specified reasons.

SUMMARY:
This is an investigator-initiated research project aimed at exploring the efficacy and safety of Adebrelimab combined with chemotherapy and Apatinib as first-line treatment for unresectable locally advanced or metastatic pulmonary neuroendocrine tumors.

This is an experimental study that has been reviewed and approved by the Ethics Committee of Beijing Chest Hospital. The study plans to enroll 39 treatment-naïve patients with unresectable locally advanced or metastatic pulmonary neuroendocrine carcinoma, who will receive first-line treatment with Adebrelimab combined with chemotherapy and Apatinib to evaluate its efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, no gender restriction;
2. Pathologically confirmed unresectable locally advanced or metastatic pulmonary neuroendocrine tumors (including large cell neuroendocrine carcinoma, small cell lung cancer, and carcinoid tumors). For carcinoid tumors, patients must be atypical carcinoid cases deemed by the investigator to require systemic treatment due to tumor-related symptoms or continuous tumor growth.
3. No prior systemic anti-tumor treatment;
4. Expected survival of at least 3 months;
5. ECOG performance status: 0-2;
6. At least one evaluable lesion based on imaging, according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1), with at least one measurable tumor lesion (non-lymph node lesion with a maximum diameter ≥ 10 mm or lymph node lesion with a short diameter ≥ 15 mm at baseline);
7. Patients with brain metastases must either be asymptomatic or have stable brain metastases to be eligible;
8. Normal function of major organs;
9. Women of childbearing potential must have used reliable contraception or have had a pregnancy test (serum or urine) within 7 days prior to enrollment, with a negative result. Both male and female patients of childbearing potential must agree to use adequate contraception during the study and for 6 months after treatment;
10. Subjects must voluntarily participate in the study, sign informed consent, demonstrate good compliance, and agree to follow-up.

Exclusion Criteria:

1. Subjects with extensive leptomeningeal metastases or active brain metastases with significant symptoms;
2. Spinal cord compression not definitively treated with surgery and/or radiotherapy, or previously diagnosed and treated spinal cord compression without clinical evidence of stabilization for at least 1 week prior to randomization;
3. Uncontrolled or symptomatic hypercalcemia;
4. Prior treatment with any T-cell co-stimulation or immune checkpoint inhibitors;
5. Use of immunosuppressive drugs within 14 days prior to the first dose of Adebrelimab;
6. Active tuberculosis (TB) within 48 weeks before screening or a history of active TB infection, regardless of prior treatment;
7. Vaccination with live attenuated or preventive vaccines within 4 weeks before the first dose or planned vaccination during the study;
8. History of allogeneic bone marrow transplantation or solid organ transplantation;
9. Severe cardiovascular disease;
10. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
11. Any active autoimmune disease or a history of autoimmune disease;
12. Coagulation abnormalities (INR > 1.5 or prothrombin time [PT] > ULN + 4 seconds or APTT > 1.5 ULN), bleeding tendency, or current thrombolytic or anticoagulation therapy;
13. Major surgery, traumatic injury, fracture, or ulcer within 4 weeks prior to enrollment, or planned major surgery during the study;
14. Severe infections such as sepsis or septic shock within 14 days before enrollment, including but not limited to hospitalization for infection, bacteremia, or severe pneumonia;
15. Significant hemoptysis within 2 months prior to enrollment, defined as more than half a teaspoon (2.5 ml) of blood daily, or any significant clinical bleeding or bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcers, baseline fecal occult blood ++ or higher, or vasculitis;
16. HBsAg positive with levels exceeding the upper limit of normal (1000 copies/ml or 500 IU/ml); patients with past or cured HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg, with normal HBV DNA during screening) may be included; HCV antibody positive with HCV viral load exceeding the upper limit of normal/HCV RNA or HCV Ab indicating acute or chronic infection; known HIV positive status or acquired immunodeficiency syndrome (AIDS);
17. Patients with a known history of allergies or suspected allergies to the study drug or any components of the study;
18. Participation in another interventional clinical trial or use of any investigational product within 4 weeks prior to signing the informed consent form (ICF);
19. History of substance abuse or inability to quit, or mental disorders;
20. History of or concurrent malignancies requiring active treatment within the past 5 years;
21. Other conditions judged by the investigator to be unsuitable for inclusion;
22. Patients with asymptomatic, stable, typical/atypical carcinoid tumors are not eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 39 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
12-month PFS rate (Progression-Free Survival rate) | 12-month

SECONDARY OUTCOMES:
Objective response rate | through study completion, an average of 2 year
Progression-free survival | through study completion, an average of 2 year
Overall survival | through study completion, an average of 2 year

IPD SHARING:
Plan to Share IPD: Undecided